CLINICAL TRIAL: NCT02217982
Title: A Pilot Study to Assess Dimethyl Fumarate (Tecfidera) Related GI Symptom Mitigation Via Food Bolus Alteration and Simethicone/Loperamide Administration
Brief Title: Pilot Study to Assess Dimethyl Fumarate Related GI Symptom Mitigation
Acronym: IIT9
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study did not meet required enrollment numbers
Sponsor: Rocky Mountain MS Research Group, LLC (Other)
Collaborators: Biogen (Industry)
Responsible Party: Principal Investigator, John F. Foley, MD, PI, Rocky Mountain MS Research Group, LLC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 009-001-TEC
Record Dates: First submitted 2014-07-30; First posted 2014-08-15 (Estimated); Results first posted 2017-01-06 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-02

CONDITIONS: Relapsing Remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Simethicone; Loperamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): Patients randomized to the standard therapy arm will be instructed to follow the normal dosing regimen for DMF with a food bolus of their choice prior to dosing. If severe symptoms (MAGIS >6.5) are noted at any time post randomization in any MAGIS category, crossover to the treatment arm will be allowed. Both groups will be asked to rate their GI symptoms over the past 24 hours using the MAGIS scale once daily.
- Treatment Arm (Active Comparator): Patients who are randomized to the treatment arm will be instructed to take 125 mg simethicone and one tablespoon of a high fat food (peanut butter)10 minutes prior to each DMF dose. If the average MAGIS score is greater than 3.5 in the diarrhea category they will also be instructed to take 2 mg loperamide three times daily.
  Interventions: Drug: Simethicone; Drug: Loperamide; Other: Peanut Butter

INTERVENTIONS:
Drug: Simethicone
  Other Names: Gas-X
  Arms: Treatment Arm
Drug: Loperamide
  Other Names: Imodium
  Arms: Treatment Arm
Other: Peanut Butter
  Arms: Treatment Arm

SUMMARY:
Single site, open label, randomized design in patients with relapsing forms of Multiple Sclerosis. At the Screening Visit, the patient will be given a diary containing the MAGIS scale to be completed once a day for the first two weeks while on Dimethyl Fumarate (DMF), including the titration period.

After two weeks or if a patient experiences 3 or more consecutive days of GI symptoms in any category of ≥3.5, the patient will return for a Baseline Visit. The MAGIS diary will be reviewed by the coordinator. Any patient who has reported an average MAGIS score of greater than or equal to 3.5 in at least one of the key categories will be randomized to a standard therapy or treatment arm. Patients who report a MAGIS of less than 3.5 during this period will be terminated from the study at this visit. Patients with an average reported MAGIS of greater than 6.5 at Baseline will be placed in the treatment arm.

Patients who are randomized to the treatment arm will be instructed to take 125 mg simethicone and one tablespoon of a high fat food (peanut butter) 10 minutes prior to each DMF dose. If the average MAGIS score is greater than 3.5 in the diarrhea category they will also be instructed to take 2 mg loperamide three times daily.

Patients randomized to the standard therapy arm will be instructed to follow the normal dosing regimen for DMF with a food bolus of their choice prior to dosing. If severe symptoms (MAGIS >6.5) are noted at any time post randomization in any MAGIS category, crossover to the treatment arm will be allowed. Both groups will be asked to rate their GI symptoms over the past 24 hours using the MAGIS scale once daily.

Both treatment arms will be observed for 6 weeks. MAGIS will be recorded once daily. Patients will return to the clinic at Week 3 and Week 6/End of Treatment for diary and compliance review. After Week 6, patients will be instructed to return to a standard therapy. MAGIS will be recorded for one more week and collected at Week 7/End of Study.

ELIGIBILITY:
Inclusion Criteria:

1. Decision to treat with DMF must precede enrollment
2. Ability to understand the purpose and risk of the study and provide authorization for the use of protected health information in accordance with the monitoring agency
3. Men or women 18 years of age or older at the time of informed consent
4. Naïve to DMF or fumaric acid esters
5. Confirmed diagnosis of a relapsing form of multiple sclerosis as verified by the Principal Investigator

Exclusion Criteria:

1. Unable to unwilling to comply with study requirements as outlined in the informed consent
2. Known active malignancies or any other major comorbidities that, in the opinion of the Investigator, would affect the outcome of the study
3. Pregnant or breastfeeding or likely to become pregnant during the course of the study. Women of child-bearing potential must practice an acceptable form of birth control
4. Previous treatment with dimethyl fumarate
5. Past history of GI malignancy, gastric ulceration refractory to medical resolution, history of gastrectomy. At the discretion of the PI, resolved GI ulceration, gastroesophageal reflux will not be exclusionary
6. Known sensitivity or allergic reaction to peanuts, simethicone, or loperamide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John F Foley, MD, Principal Investigator — Rocky Mountain MS Research Group
Locations (1):
- Rocky Mountain MS Research Group, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Arm: Patients who are randomized to the treatment arm will be instructed to take 125 mg simethicone and one tablespoon of a high fat food (peanut butter)10 minutes prior to each DMF dose. If the average MAGIS score is greater than 3.5 in the diarrhea category they will also be instructed to take 2 mg loperamide three times daily.
  Simethicone
  Loperamide
  Peanut Butter
Period: Overall Study
Arm/Group | Control Group | Treatment Arm
Started | 1 | 4
Completed | 0 (Trial closed before patient finished) | 3
Not Completed | 1 | 1
Not completed — Trial discontinued | 1 | 0
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: 5 patients total qualified for the trial after monitoring of GI symptoms after initiation of DMF
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Treatment Arm | Total
Number analyzed (Participants) | 1 | 4 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 4 | 5
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Reported GI Symptoms
Description: The primary endpoint will be severity of GI events as measured by the MAGIS scale for subjects in the treatment arm compared to the standard therapy arm.
Time Frame: 7 Weeks
Population: Trial was shut down early as not enough patients qualified with GI symptoms their first 2 weeks after initiating DMF therapy
Arm/Group | Control Group | Treatment Arm
Number analyzed (Participants) | 0 | 0
Value | 0 | 0

2. Secondary Outcome: Diarrhea Reduction
Description: The secondary objective is to assess the reduction in diarrhea in the treatment group compared to the control.
Time Frame: 7 Weeks
Population: Not enough patients qualified and the study was terminated early.
Arm/Group | Control Group | Treatment Arm
Number analyzed (Participants) | 0 | 0
Value | 0 | 0

3. Other Pre Specified Outcome: Number of Participants With Pre-Existing GI Conditions
Description: The tertiary objective is to gather further data regarding pre-existing conditions (GE reflex, gastric bypass, stomach ulcer, etc) and their possible relationship to GI symptoms when initiating DMF.
Time Frame: 7 Weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: approximately 10 weeks from consent to end of study
Arm/Group | Control Group | Treatment Arm
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/4
Other Adverse Events (participants affected / at risk) | 0/1 | 0/4

LIMITATIONS AND CAVEATS:
This trial was closed down early because the anticipated number of patients experiencing GI symptoms was not met - therefore not enough patients qualified for the treatment and control arms for analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes